CLINICAL TRIAL: NCT02715856
Title: Using Telemonitoring to Optimize the Mobility of Cancer Survivors With Skeletal Metastases After Surgery to Preserve Limb Function
Brief Title: Telemonitoring After Surgery to Preserve Limb Function in Optimizing Mobility in Cancer Survivors With Skeletal Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to software issues and depletion of funds the protocol was terminated early
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-0966; NCI-2016-00544 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0966 (Other: M D Anderson Cancer Center); 2015-00051255-Y1 (Other Grant/Funding Number: Cancer Survivorship Research Seed Money Grant)
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Bone Metastases; Cancer Survivor; Metastatic Malignant Neoplasm in the Bone
Keywords: Bone metastases; Intramedullary nailing surgery; IM; Physical tasks; Surveys; Questionnaires; Smartphone; Tablet; Telemedicine; Telemonitoring
MeSH Terms: interventions — Continuous Glucose Monitoring; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (standard follow up, physical activity measurement) (Active Comparator): Patients undergo standard face-to-face follow up visits at 2, 6, 12, and 24 weeks after surgery. Patients also undergo a physical activity assessment over 15 minutes.
  Interventions: Other: Physical Activity Measurement; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Standard Follow-Up Care; Other: Survey Administration
- Group II (mobile surveillance) (Experimental): Patients undergo standard face-to-face follow up visits as in Group I. Patients also undergo mobile surveillance comprising use of a mobile device application to send photos and videos to study staff and engage in video conferences at 3, 7, 13, and 25 weeks after surgery.
  Interventions: Other: Monitoring Device; Other: Physical Activity Measurement; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Standard Follow-Up Care; Other: Survey Administration

INTERVENTIONS:
Other: Monitoring Device — Undergo surgical wound and physical activity monitoring
  Other Names: Monitor
  Arms: Group II (mobile surveillance)
Other: Physical Activity Measurement — Undergo physical activity measurement
  Other Names: Activity
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Standard Follow-Up Care — Undergo standard follow-up care
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized pilot trial studies telemonitoring after surgery to preserve limb function in optimizing mobility in cancer survivors with cancer spread to the bone. The use of mobile devices for telemonitoring may improve the delivery of cost-effective, high-quality, standardized surveillance of cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and evaluate the feasibility of a method that enhances surveillance in cancer survivors by using mobile devices in addition to face-to-face visits following surgery for bone metastases.

SECONDARY OBJECTIVES:

I. To evaluate how well the face-to-face follow-up format can be adapted to using mobile devices for remote surveillance.

II. Limited efficacy testing of the remote surveillance program. III. To obtain information on acceptability of the mobile surveillance format by patients and clinicians.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (CONTROL): Patients undergo standard face-to-face follow up visits at 2, 6, 12, and 24 weeks after surgery. Patients also undergo a physical activity assessment over 15 minutes.

GROUP II (MOBILE SURVEILLANCE): Patients undergo standard face-to-face follow up visits as in Group I. Patients also undergo mobile surveillance comprising use of a mobile device application to send photos and videos to study staff and engage in video conferences at 3, 7, 13, and 25 weeks after surgery.

After completion of study, patients are followed up at 24-25 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been scheduled for an intramedullary nailing (IM) surgery with the department of Orthopaedic Oncology at University of Texas (UT) MD Anderson Cancer Center
* Are able to read and write English 3) Are 18 years or older
* Are willing and able to use a smartphone or tablet comfortably
* Have access to mobile hot spot, wireless internet, and/or cellular service
* Must have a caregiver or assistance at home who can assist with collecting physical therapy (PT) measures

Exclusion:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Satcher, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I (Control): Patients undergo standard face-to-face follow up visits at 2, 6, 12, and 24 weeks after surgery. Patients also undergo a physical activity assessment over 15 minutes.
  Physical Activity Measurement: Undergo physical activity measurement
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Standard Follow-Up Care: Undergo standard follow-up care
  Survey Administration: Ancillary studies
- Phase II (Mobile Surveillance): Patients undergo standard face-to-face follow up visits as in Group I. Patients also undergo mobile surveillance comprising use of a mobile device application to send photos and videos to study staff and engage in video conferences at 3, 7, 13, and 25 weeks after surgery.
  Monitoring Device: Undergo surgical wound and physical activity monitoring
  Physical Activity Measurement: Undergo physical activity measurement
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Standard Follow-Up Care: Undergo standard follow-up care
  Survey Administration: Ancillary studies
Period: Overall Study
Arm/Group | Phase I (Control) | Phase II (Mobile Surveillance)
Started | 18 | 52
Completed | 0 | 0
Not Completed | 18 | 52
Not completed — Software Issues | 12 | 7
Not completed — Death | 6 | 5
Not completed — Non- Compliant | 0 | 40

BASELINE CHARACTERISTICS:
Groups:
- Phase I (Standard Follow up, Physical Activity Measurement): Patients undergo standard face-to-face follow up visits at 2, 6, 12, and 24 weeks after surgery. Patients also undergo a physical activity assessment over 15 minutes.
  Physical Activity Measurement: Undergo physical activity measurement
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Standard Follow-Up Care: Undergo standard follow-up care
  Survey Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Phase I (Standard Follow up, Physical Activity Measurement) | Phase II (Mobile Surveillance) | Total
Number analyzed (Participants) | 18 | 52 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 59 (13) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 30 | 40
  Male | 8 | 22 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 52 | 70

OUTCOME MEASURES:

1. Primary Outcome: Inter-Rater Agreement on the Physician Assessed Score
Description: Inter-rater agreement on the physician assessed score defined as less than 10% difference between the Musculoskeletal Tumor Society (MSTS) scores evaluated using video vs. face-to-face follow ups.
Time Frame: 7 months
Population: Due to software issues and depletion of funds the protocol was terminated early and the participants did not complete assessments per protocol at given point, no data collected.
Arm/Group | Phase I (Standard Follow up, Physical Activity Measurement) | Phase II (Mobile Surveillance)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Completion of Follow-Up Assessments
Description: Participant considered having completed the follow-up assessments if the three outcomes are documented for the 2-, 6-, 12, and 24-week evaluations. Follow-up assessment information taken from Musculoskeletal Tumor Society Scores (MSTS), Timed "Up and Go" test (TUG), and Patient Reported Outcomes Measurement Information System (PROMIS).
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Phase I (Standard Follow up, Physical Activity Measurement) | Phase II (Mobile Surveillance)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Phase I (Standard Follow up, Physical Activity Measurement) | Phase II (Mobile Surveillance)
All-Cause Mortality (participants affected / at risk) | 6/18 | 5/52
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/52
Other Adverse Events (participants affected / at risk) | 0/18 | 0/52

LIMITATIONS AND CAVEATS:
Due to software issues and depletion of funds the protocol was terminated early and the participants did not complete assessments per protocol at given point, no data collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT02715856/Prot_SAP_000.pdf